CLINICAL TRIAL: NCT05701072
Title: Development of a Screening Tool for Difficult Embryo Transfers
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Mustafa Baris Ata, Principal Investigator, ART Fertility Clinics LLC
Other Study IDs: 2208-ABU-007-BA
Record Dates: First submitted 2023-01-17; First posted 2023-01-27 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Infertility
Keywords: infertility; embryo transfer
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All participants
  Interventions: Procedure: Oocyte Pick Up; Procedure: Embryo Transfer

INTERVENTIONS:
Procedure: Oocyte Pick Up — The screening questionnaire will be filled by the Physician doing the OPU. The screening questionnaire will be informed by the participant's history. Cervix will be visualized during routine vaginal cleansing for OPU, and its appearance (size, and deviation) will be recorded in the screening questionnaire after the OPU procedure. Finally, a screenshot of the ultrasound used for OPU, showing the cervix and cervical canal in the sagittal plane will be taken during routine procedure and saved in electronic chart.
Procedure: Embryo Transfer — When the participants comes back for ET during her routine treatment, ET will be done in exactly the same way in routine treatment. Participant will not undergo any additional manipulation, intervention, nor the procedure will take longer. The Embryologist assisting the procedure will record the duration of the procedure, from the moment the Physician takes the outer ET catheter to his/her hand until he/she passes the cervix and calls for the inner catheter loaded with the embryo. Up on completion of the ET procedure as routine practice, the Physician will fill a questionnaire about the procedure.

SUMMARY:
This study aims to investigate the accuracy of a proposed screening tool in identifying difficult embryo transfers (ETs) without doing a mock ET.

DETAILED DESCRIPTION:
So far there has never been a screening tool to identify difficult ETs without doing a mock ET. This is a prospective, longitudinal study including at least 200 ETs. All women undergo a speculum examination at the time of transvaginal oocyte pick-up (OPU), the screening questionnaire will be filled by the Physician doing the OPU procedure. On the day of real ET, the Physician doing the ET will be blinded for the screening result, and fill a second questionnaire after the ET. Combined with the Embryologist recorded parameters, this second questionnaire will be used to categorize ETs as difficult or normal. Participants will NOT undergo any procedures beyond their routine treatment. Once the targeted number of participants are recruited, the questionnaires will be matched to see the accuracy of the screening questionnaire to identify difficult ETs.

Identification of difficult ETs with a non-invasive, free of cost questionnaire can enable selective mock transfers and facilitate the real ET for patients, who would otherwise be only recognized on the day of real ET, after their embryos have been already thawed for transfer.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing an ET is eligible.

Exclusion Criteria:

* No exclusion criteria, women can participate with multiple ET procedures.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: All women undergoing an ET in ART Fertility Clinics Abu Dhabi and Dubai.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of difficult ET | Approximately 4 months
Percentage of screening questionnaires suggesting a difficult ET | Approximately 4 months
Accuracy of the screening tool to predict difficult ET | Approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Study Director — ART Fertility Clinics LLC
Locations (2):
- United Arab Emirates (2):
  - ART Fertility Clinics LLC, Abu Dhabi, Abu Dhabi Emirate
  - ART Fertility Clinics LLC, Dubai

REFERENCES:
- [Background] Cirillo F, Patrizio P, Baccini M, Morenghi E, Ronchetti C, Cafaro L, Zannoni E, Baggiani A, Levi-Setti PE. The human factor: does the operator performing the embryo transfer significantly impact the cycle outcome? Hum Reprod. 2020 Feb 29;35(2):275-282. doi: 10.1093/humrep/dez290. PMID 32100020
- [Background] Dessolle L, Freour T, Barriere P, Jean M, Ravel C, Darai E, Biau DJ. How soon can I be proficient in embryo transfer? Lessons from the cumulative summation test for learning curve (LC-CUSUM). Hum Reprod. 2010 Feb;25(2):380-6. doi: 10.1093/humrep/dep391. Epub 2009 Nov 18. PMID 19923166
- [Background] Lopez MJ, Garcia D, Rodriguez A, Colodron M, Vassena R, Vernaeve V. Individualized embryo transfer training: timing and performance. Hum Reprod. 2014 Jul;29(7):1432-7. doi: 10.1093/humrep/deu080. Epub 2014 Apr 29. PMID 24781427
- [Background] Noyes N, Licciardi F, Grifo J, Krey L, Berkeley A. In vitro fertilization outcome relative to embryo transfer difficulty: a novel approach to the forbidding cervix. Fertil Steril. 1999 Aug;72(2):261-5. doi: 10.1016/s0015-0282(99)00235-6. PMID 10438992
- [Background] Kably Ambe A, Campos Canas JA, Aguirre Ramos G, Carballo Mondragon E, Carrera Lomas E, Ortiz Reyes H, Kisel Laska R. [Evaluation of two transfer embryo systems performed by six physicians]. Ginecol Obstet Mex. 2011 Apr;79(4):196-9. Spanish. PMID 21966806
- [Background] Wood MA, Kerrigan KL, Burns MK, Glenn TL, Ludwin A, Christianson MS, Bhagavath B, Lindheim SR. Overcoming the Challenging Cervix: Identification and Techniques to Access the Uterine Cavity. Obstet Gynecol Surv. 2018 Nov;73(11):641-649. doi: 10.1097/OGX.0000000000000614. PMID 30468239
- [Derived] Ata B, Lawrenz B, Melado L, Del Gallego R, Coughlan C, Ruiz F, Marqueta Marques L, El-Damen A, Elkhatib I, Fatemi HM. The ART-ET screening tool: an easy-to-use non-invasive screening method to predict difficult embryo transfers in advance. Hum Reprod. 2025 Apr 1;40(4):647-653. doi: 10.1093/humrep/deaf002. PMID 39938557